CLINICAL TRIAL: NCT04042792
Title: Characterization of Adalimumab Concentrations in Pediatric Patients With Inflammatory Rheumatic Disease With and Without Methotrexate (ADA in PiRD)
Brief Title: Characterization of Adalimumab Concentrations in Pediatric Patients With Inflammatory Rheumatic Disease With and Without Methotrexate
Acronym: ADA in PiRD
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00916; ks18Pfister2
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Rheumatic Diseases
Keywords: pharmacokinetics; pharmacodynamics; Adalimumab; methotrexate; drug-drug interaction; trough ADA concentration; peak ADA concentration; Pediatric inflammatory rheumatic diseases
MeSH Terms: conditions — Rheumatic Diseases | interventions — Pharmacokinetics; Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADA for ≥12 weeks and concomitant MTX therapy: PiRD patients with ADA for ≥12 weeks and concomitant MTX therapy (oral or subcutaneous)
  Interventions: Other: pharmacokinetics (PK) measurement
- ADA for ≥ 12 weeks without MTX: PiRD patients with ADA for ≥ 12 weeks without MTX ≥ 12 weeks (or never exposed to MTX)
  Interventions: Other: pharmacokinetics (PK) measurement

INTERVENTIONS:
Other: pharmacokinetics (PK) measurement — two ADA-PK samples will be collected during routine rheumatology visits in case of medical indicated blood draw (1 trough PK sample and 1 random PK sample per subject)

SUMMARY:
This study is to assess standardized Adalimumab (ADA) concentrations in Pediatric inflammatory rheumatic diseases (PiRD) patients treated with ADA for ≥ 12 weeks with and without concomitant methotrexate (MTX) therapy and to assess peak and trough ADA concentrations in ADA naïve patients after first ADA administration with and without MTX (pre-phase).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of a juvenile idiopathic Arthritis (JIA), uveitis or chronic recurrent multifocal osteomyelitis (CRMO)
* Medical indication for initiation of ADA treatment or established ADA therapy for ≥ 12 weeks
* Exclusion of chronic infections
* No parallel treatment with other biologic medications
* Available patient history since ADA start
* No pregnancy
* Ability to comply with the entire study protocol
* Willingness to participate with signed informed consent

Exclusion Criteria:

* Other rheumatic inflammatory diseases
* Age < 2 years or >18 years
* PiRD patients and parents with cognitive impairments preventing to understand study requirements
* Additional severe chronic disease (kidney failure, liver insufficiency), malignancies or prior chemotherapy

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: PiRD patients treated with ADA for medical reasons at the University Children's Hospital Basel/ Switzerland and at the University Children's Hospital of Tuebingen/ Germany
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
ADA concentration (in mg/L) | at study inclusion
  ADA concentration (in mg/L)
ADA concentration (in mg/L) | during regular clinical follow up 3-6 months after inclusion
  ADA concentration (in mg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Pfister, Prof. Dr., Principal Investigator — University Children's Hospital Basel (UKBB), University of Basel
Locations (2):
- University Children's Hospital Tubingen, Tübingen, Germany
- University of Basel Children's Hospital, Basel, Switzerland

REFERENCES:
- [Derived] Welzel T, Golhen K, Atkinson A, Gotta V, Ternant D, Kuemmerle-Deschner JB, Michler C, Koch G, van den Anker JN, Pfister M, Woerner A. Prospective study to characterize adalimumab exposure in pediatric patients with rheumatic diseases. Pediatr Rheumatol Online J. 2024 Jan 2;22(1):5. doi: 10.1186/s12969-023-00930-8. PMID 38167019